CLINICAL TRIAL: NCT00192647
Title: A Phase IV, Randomised, Multicentre, Efficacy and Safety Study Examining the Effect of Induction Dosing With the Combination of Peginterferon Alfa-2a and Ribavirin in Patients With Chronic Hepatitis C Infected With Hepatitis C Genotype 1
Brief Title: A Study of Induction Dosing With Peginterferon Alfa-2a and Ribavirin in Participants With Chronic Hepatitis C (CHC) Genotype 1 Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17908
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

ARMS (2):
- PEG-IFN alfa-2a+Ribavirin - Induction Treatment (Experimental): Participants will receive 12 weeks of induction therapy with PEG-IFN alfa-2a (Pegasys), 360 micrograms (mcg) subcutaneous (SC) once weekly, along with ribavirin, 1000 or 1200 milligrams (mg) orally daily in divided doses. Thereafter, the dose of PEG-IFN alfa-2a will be reduced to 180 mcg SC once weekly and the ribavirin dose maintained for the remaining 36 weeks of treatment.
  Interventions: Drug: PEG-IFN alfa-2a; Drug: Ribavirin
- PEG-IFN alfa-2a+Ribavirin - Standard Treatment (Experimental): Participants will receive 48 weeks of standard therapy with PEG-IFN alfa-2a, 180 mcg SC once weekly, along with ribavirin, 1000 or 1200 mg orally daily in divided doses.
  Interventions: Drug: PEG-IFN alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: PEG-IFN alfa-2a — PEG-IFN alfa-2a will be administered once weekly for 48 weeks, at doses specified in respective arms.
  Other Names: Pegasys
Drug: Ribavirin — Ribavirin 1000 or 1200 mg orally daily in divided doses, with the dose determined based on body weight, for 48 weeks.
  Other Names: Copegus

SUMMARY:
This study will evaluate the addition of a higher-dose induction treatment period with peginterferon (PEG-IFN) alfa-2a (Pegasys) and ribavirin prior to standard-dose treatment with PEG-IFN alfa-2a and ribavirin, compared to standard-dose treatment, in treatment-naive participants with CHC, genotype 1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic CHC, genotype 1
* Chronic liver disease consistent with CHC on a biopsy sample obtained within the previous 36 months as judged by a local pathologist (all countries except Australia)
* Infection with Hepatitis C virus (Australian sites only had to meet Section 100 criteria for treatment with PEG-IFN alfa-2a plus ribavirin)
* Compensated liver disease
* Naive to interferon-based therapy for CHC infection

Exclusion Criteria:

* Systemic antiviral, antineoplastic, or immunomodulatory treatment within 6 months of study drug
* Coinfection with active hepatitis A or B virus, or with human immunodeficiency virus (HIV)
* Chronic liver disease other than CHC infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2004-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (40):
- Argentina (3):
  - Buenos Aires
  - La Plata
  - Rosario
- Australia (25):
  - Adelaide
  - Bankstown
  - Box Hill
  - Brisbane
  - Cottontree
  - Darlinghurst
  - Douglas
  - Fitzroy
  - Fremantle
  - Geelong
  - Greenslopes
  - Kingswood
  - Lismore
  - Liverpool
  - Melbourne
  - Miranda
  - Nedlands
  - New Lambton Heights
  - Parkville
  - Perth
  - Sydney
  - Victoria
  - Woden
  - Wollongong
  - Woolloongabba
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Mississauga, Ontario
  - Montreal, Quebec
- Mexico (2):
  - Guadalajara
  - Monterrey
- New Zealand (3):
  - Auckland
  - Hamilton
  - Riccarton, Christchurch
- Thailand (2):
  - Bangkok
  - Chiang Mai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of total 896 randomized participants, 25 participants (15 in the induction group and 10 in the standard group) did not receive study drug.
Groups:
- PEG-IFN Alfa-2a+Ribavirin - Induction Treatment: Participants received 12 weeks of induction therapy with peginterferon (PEG-IFN) alfa-2a (Pegasys), 360 micrograms (mcg) subcutaneous (SC) once weekly, along with ribavirin, 1000 or 1200 milligrams (mg) orally daily in divided doses, with the dose determined based on body weight. Thereafter, the dose of PEG-IFN alfa-2a was reduced to 180 mcg SC once weekly and the ribavirin dose was maintained for the next 36 weeks of treatment.
- PEG-IFN Alfa-2a+Ribavirin - Standard Treatment: Participants received 48 weeks of standard therapy with PEG-IFN alfa-2a, 180 mcg SC once weekly, along with ribavirin, 1000 or 1200 mg orally daily in divided doses, with the dose determined based on body weight.
Period: Overall Study
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment
Started | 448 | 448
Treated | 433 | 438
Completed | 320 | 302
Not Completed | 128 | 146
Not completed — Death | 1 | 1
Not completed — Adverse Event | 35 | 29
Not completed — Laboratory Test Abnormality | 4 | 2
Not completed — Insufficient Therapeutic Response | 53 | 83
Not completed — Entry Criteria Violation | 6 | 6
Not completed — Protocol Violation | 3 | 1
Not completed — Refused Treatment/Did not Cooperate | 10 | 8
Not completed — Failure to Return | 11 | 13
Not completed — Other/Administrative | 5 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis population included all randomized participants who received at least 1 dose of study drug.
Groups:
- PEG-IFN Alfa-2a+Ribavirin - Induction Treatment: Participants received 12 weeks of induction therapy with PEG-IFN alfa-2a, 360 mcg SC once weekly, along with ribavirin, 1000 or 1200 mg orally daily in divided doses, with the dose determined based on body weight. Thereafter, the dose of PEG-IFN alfa-2a was reduced to 180 mcg SC once weekly and the ribavirin dose was maintained for the next 36 weeks of treatment.
- Total: Total of all reporting groups
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment | Total
Number analyzed (Participants) | 433 | 438 | 871
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9.55) | 43.3 (9.19) | 43.4 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 153 | 288
  Male | 298 | 285 | 583

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response According to Scheduled Treatment Period
Description: Sustained virological response was calculated as the percentage of participants with undetectable (less than [<] 15 international units per milliliter [IU/mL]) hepatitis C virus (HCV) ribonucleic acid (RNA) as measured by the Roche TaqMan HCV Test 24 weeks after completion of the scheduled 48-week treatment period.
Time Frame: Week 72
Population: ITT analysis population
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment
Number analyzed (Participants) | 433 | 438
percentage of participants | 53 | 50
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a+Ribavirin - Induction Treatment vs PEG-IFN Alfa-2a+Ribavirin - Standard Treatment; Test type: Superiority or Other; p = 0.2893, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by viral load and country; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.88 to 1.52]

2. Secondary Outcome: Percentage of Participants With End-of-Treatment Virological Response According to Scheduled Treatment Period
Description: Virological response at the end of the scheduled treatment period was defined as the percentage of participants with undetectable (<15 IU/mL) HCV RNA as measured by the Roche TaqMan HCV Test at Week 48.
Time Frame: Weeks 48
Population: ITT analysis population
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment
Number analyzed (Participants) | 433 | 438
percentage of participants | 70 | 66
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a+Ribavirin - Induction Treatment vs PEG-IFN Alfa-2a+Ribavirin - Standard Treatment; Test type: Superiority or Other; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.91 to 1.63]

3. Secondary Outcome: Percentage of Participants With Virological Responses Over Time
Description: Virological response was defined as undetectable HCV RNA (<15 IU/mL) as measured by the Roche TaqMan HCV Test. Participants without HCV RNA measurements at a study week are considered non responders at that study week.
Time Frame: Weeks 4, 8, 12, and 24
Population: ITT analysis population
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment
Number analyzed (Participants) | 433 | 438
percentage of participants
  Week 4 | 36.0 | 26.3
  Week 8 | 60.5 | 49.8
  Week 12 | 74.4 | 61.6
  Week 24 | 75.1 | 67.8
Statistical Analysis 1: Comparison: PEG-IFN Alfa-2a+Ribavirin - Induction Treatment vs PEG-IFN Alfa-2a+Ribavirin - Standard Treatment; Week 4; Test type: Superiority or Other; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.24 to 2.27]
Statistical Analysis 2: Comparison: PEG-IFN Alfa-2a+Ribavirin - Induction Treatment vs PEG-IFN Alfa-2a+Ribavirin - Standard Treatment; Week 8; Test type: Superiority or Other; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.24 to 2.17]
Statistical Analysis 3: Comparison: PEG-IFN Alfa-2a+Ribavirin - Induction Treatment vs PEG-IFN Alfa-2a+Ribavirin - Standard Treatment; Week 12; Test type: Superiority or Other; Odds Ratio (OR) = 1.88, 95% CI 2-sided [1.40 to 2.53]
Statistical Analysis 4: Comparison: PEG-IFN Alfa-2a+Ribavirin - Induction Treatment vs PEG-IFN Alfa-2a+Ribavirin - Standard Treatment; Week 24; Test type: Superiority or Other; Odds Ratio (OR) = 1.46, 95% CI 2-sided [1.08 to 1.98]

4. Secondary Outcome: Percentage of Participants With Relapse of End-of-treatment Virological Response
Description: Relapse was determined based on virological response at the actual end of treatment and was calculated by dividing the number of participants who achieved a virological response at end of treatment but later had detectable HCV RNA at the last assessment post-treatment by the number of participants with a virological response at end of treatment, defined as undetectable HCV RNA (<15 IU/mL). Participants who achieved a virological response at end of treatment but did not have any HCV RNA assessment during follow-up were excluded and were not considered as having relapsed. However, if no assessment was available within the end of-treatment time window but the participant had a sustained virological response according to the actual treatment period, backward imputation was used and the participant was considered to have achieved an end-of-treatment virological response in the analysis.
Time Frame: Actual end of treatment (Week 48) up to last follow up (maximum up to Week 72)
Population: ITT analysis population. Here, number of participants analyzed signifies participants who had end of treatment virologic response and had HCV RNA measurement available during follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment
Number analyzed (Participants) | 297 | 280
percentage of participants | 24 | 22

5. Secondary Outcome: Percentage of Participants With Predictive Values of Virological Response for Sustained Virological Response
Description: The ability of virological responses to predict sustained virological response according to the scheduled treatment periods was assessed in terms of positive predictive value (PPV) and negative predictive value (NPV). The PPV indicates probability of achievement of viral suppression (undetectable HCV RNA) for achieving a sustained virological response and the NPV indicates probability of not achieving viral suppression for not achieving a sustained virological response. The PPV at Week 4 or 12 was calculated as the number of participants who achieved viral suppression both at Week 4 or 12 and at Week 72 divided by the number of participants who achieved viral suppression at Week 4 or 12, multiplied by 100. The NPV at Week 4 or 12 was calculated as the number of participants who failed to achieve viral suppression at Week 4 or 12 and at Week 72 divided by the number of participants who failed to achieve viral suppression at Week 4 or 12, multiplied by 100.
Time Frame: Weeks 4, 12, and 72
Population: ITT analysis population; participants who did not have an HCV RNA measurement at Week 4 or 12 and at Week 72 were excluded from the analysis. Here, number of participants analyzed = number of participants evaluable for this outcome measure; 'n' = number of participants analyzed at specified time point for reported group, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment
Number analyzed (Participants) | 416 | 419
percentage of participants
  Week 4: PPV (n= 416, 419) | 76 | 80
  Week 4: NPV (n= 416, 419) | 60 | 60
  Week 12: PPV (n= 412, 413) | 66 | 72
  Week 12: NPV (n= 412, 413) | 87 | 87

6. Secondary Outcome: Change From Baseline in Log10 HCV RNA Values
Description: The mean decrease in log10 HCV RNA levels from baseline was assessed in both the induction group and the standard group.
Time Frame: Baseline, Weeks 4, 8, 12, 24, and at end of treatment (EoT) (maximum up to Week 48)
Population: ITT analysis population; Here, number of participants analyzed = number of participants evaluable for this outcome measure; 'n' = number of participants analyzed at specified time point for reported group, respectively.
Measure: Mean (Standard Deviation); unit: Log 10 IU/mL
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment
Number analyzed (Participants) | 427 | 431
Log 10 IU/mL
  Baseline (n=427,431) | 6.19 (0.72) | 6.17 (0.76)
  Change at Week 4 (n=410,412) | -3.42 (1.59) | -2.75 (1.71)
  Change at Week 8 (n=399,406) | -4.26 (1.36) | -3.68 (1.72)
  Change at Week 12 (n=406,407) | -4.57 (1.21) | -4.04 (1.67)
  Change at Week 24 (n=369,369) | -4.58 (1.37) | -4.28 (1.70)
  Change at EoT (n=425,426) | -4.49 (1.44) | -4.13 (1.76)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 72
Description: Safety analysis population included all participants who received at least 1 injection of PEG-IFN alfa-2a or 1 dose of ribavirin and had at least 1 post-baseline safety assessment.
Arm/Group | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment
Serious Adverse Events (participants affected / at risk) | 46/433 | 45/438
Other Adverse Events (participants affected / at risk) | 428/433 | 430/438
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment (N=433) | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment (N=438)
Pneumonia (Infections and infestations) | 4 | 1
Appendicitis (Infections and infestations) | 3 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bartholin's abscess (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 3
Suicide attempt (Psychiatric disorders) | 1 | 3
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression suicidal (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 6 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1
Chest pain (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Optic Ischaemic Neuropathy (Eye disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hypotonic urinary bladder (Renal and urinary disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Finger amputation (Surgical and medical procedures) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN Alfa-2a+Ribavirin - Induction Treatment (N=433) | PEG-IFN Alfa-2a+Ribavirin - Standard Treatment (N=438)
Anaemia (Blood and lymphatic system disorders) | 45 | 39
Neutropenia (Blood and lymphatic system disorders) | 57 | 43
Dry eye (Eye disorders) | 32 | 25
Vision blurred (Eye disorders) | 44 | 39
Abdominal pain (Gastrointestinal disorders) | 37 | 31
Constipation (Gastrointestinal disorders) | 22 | 39
Diarrhoea (Gastrointestinal disorders) | 100 | 76
Dry mouth (Gastrointestinal disorders) | 54 | 44
Mouth ulceration (Gastrointestinal disorders) | 43 | 46
Nausea (Gastrointestinal disorders) | 178 | 168
Vomiting (Gastrointestinal disorders) | 49 | 48
Asthenia (General disorders) | 26 | 17
Chills (General disorders) | 64 | 34
Fatigue (General disorders) | 159 | 174
Influenza like illness (General disorders) | 180 | 183
Injection site erythema (General disorders) | 44 | 46
Injection site reaction (General disorders) | 25 | 23
Irritability (General disorders) | 109 | 111
Pyrexia (General disorders) | 66 | 47
Lower respiratory tract infection (Infections and infestations) | 24 | 15
Weight decreased (Investigations) | 120 | 87
Decreased appetite (Metabolism and nutrition disorders) | 160 | 113
Arthralgia (Musculoskeletal and connective tissue disorders) | 82 | 76
Back pain (Musculoskeletal and connective tissue disorders) | 44 | 39
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 114 | 97
Disturbance in attention (Nervous system disorders) | 38 | 46
Dizziness (Nervous system disorders) | 84 | 79
Dysgeusia (Nervous system disorders) | 36 | 31
Headache (Nervous system disorders) | 227 | 208
Lethargy (Nervous system disorders) | 134 | 123
Memory impairment (Nervous system disorders) | 23 | 33
Anxiety (Psychiatric disorders) | 46 | 43
Depressed mood (Psychiatric disorders) | 18 | 24
Depression (Psychiatric disorders) | 83 | 82
Insomnia (Psychiatric disorders) | 195 | 208
Mood altered (Psychiatric disorders) | 25 | 21
Mood swings (Psychiatric disorders) | 32 | 41
Cough (Respiratory, thoracic and mediastinal disorders) | 70 | 61
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 41
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 48 | 30
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26 | 19
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 28 | 29
Alopecia (Skin and subcutaneous tissue disorders) | 122 | 99
Dry skin (Skin and subcutaneous tissue disorders) | 76 | 86
Pruritus (Skin and subcutaneous tissue disorders) | 76 | 88
Rash (Skin and subcutaneous tissue disorders) | 110 | 116
Rash pruritic (Skin and subcutaneous tissue disorders) | 24 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.